CLINICAL TRIAL: NCT01310387
Title: A Randomized Prospective Controlled Study of Active Pain Management in Lung Cancer Outpatients (APM)
Brief Title: Prospective Study of Active Pain Management in Lung Cancer Outpatients (APM)
Acronym: APM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Principal Investigator, Young-Chul Kim, Professor, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PAIN_LCA_2011
Record Dates: First submitted 2011-02-01; First posted 2011-03-08 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Cancer pain; Opioid
MeSH Terms: conditions — Lung Neoplasms; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- active pain management (Experimental): active pain management (APM) by specialized nurses for cancer pain
  Interventions: Behavioral: Active pain management

INTERVENTIONS:
Behavioral: Active pain management — Active pain management will be provided by specialized pain nurse, such as telephone counseling for toxicity control and opioid dose modification.

SUMMARY:
This study is:

* A single-center, randomized, prospective controlled trial.
* To prove superiority of active pain management group compared to control group by the percent of pain intensity difference of outpatients with lung cancer pain.
* 204 patients will be recruited.

DETAILED DESCRIPTION:
* The recruited patients in both group will be provided the education about pain-killer, and received medicines including opioids according to their numeric rating scale (NRS)
* Active management group will be provided additional telephone counseling and dosage modification by specialized nurse for cancer pain.
* The percent of pain intensity difference (%PID)

  * PID = (NRS of visit 1 - NRS of visit 3)/NRS of visit 1

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with lung cancer.
* The patients with uncontrolled lung cancer pain - more than and equal NRS 4 pain during previous 24 hours for background pain, or more than and equal 3 times/day for breakthrough painkiller medication.
* Over 20 year-old male or female.
* The patients can be able to received telephone counseling by investigator's decision.

Exclusion Criteria:

* Drug or alcohol abusers.
* Child-bearing women or pregnant women.
* The patients with moderate to severe psychiatric problems.
* The patients who have hypersensitivity to opioids.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The percent of pain intensity difference | visit 3 (6 to 8 weeks)
  The percent of pain intensity difference (%PID)
  %PID = (NRS of visit 1 - NRS of visit 3)/NRS of visit 1

SECONDARY OUTCOMES:
Patients' satisfaction score about pain management | visit 3 (6 to 8 weeks)
  Qustionnaire of 5-point scale
Eastern Cooperative Oncology Group (ECOG) Performance score | visit 3 (6 to 8 weeks)
  ECOG performance status: 0,1,2,3,4
Assessment of Korean Brief Pain Inventory score | visit 3 (6 to 8 weeks)
  Qustionnaire; K-BPI(Korean Brief Pain Inventory)
Investigator's global assessment score | visit 3 (6 to 8 weeks)
  Qustionnaire of 5-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Kim, MD,PhD, Study Chair — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Jeonnam, South Korea